CLINICAL TRIAL: NCT04083742
Title: The Heidelberg Engineering ANTERION Anterior Segment Metrics Precision and Agreement Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B-2018-3
Record Dates: First submitted 2019-08-23; First posted 2019-09-10 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Narrow Angle; Open Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Eyes with Open Angle: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION
- Eyes with Narrow Angle: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION

INTERVENTIONS:
Device: ANTERION — 3 repeat angle measurements performed on each of the 3 Anterion devices and the 3 reference devices

SUMMARY:
This is a prospective clinical study that will be conducted at one clinical site located in the United States to assess anterior segment metrics with the ANTERION

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 years or older
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions
3. Able to fixate
4. With at least one of following eye status for the corresponding eye population:

A. Eye with Open Angle (defined by Spaeth gonioscopy grading)

B. Eye with Narrow Angle (defined by Spaeth gonioscopy grading)

Exclusion Criteria:

1. Subjects which were enrolled in the B-2018-1 study
2. Active infection or inflammation in either eye
3. Insufficient tear film or corneal reflex
4. Physical inability to be properly positioned at the study devices or eye exam equipment
5. Rigid contact lens wear during 2 weeks prior to day when study device acquisitions take place
6. Soft lenses worn within one hour prior to study device acquisitions

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eyes with narrow angle and eyes with open angle
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Repeatability and Reproducibility 1 | 1 day
  Reproducibility and repeatability of Spur to Spur distance parameter [mm] of ANTERION and the reference device
Repeatability and Reproducibility 2 | 1 day
  Reproducibility and repeatability of Angle to Angle distance parameter [mm] of ANTERION and the reference device
Repeatability and Reproducibility 3 | 1 day
  Reproducibility and repeatability of Lens Vault parameter [µm] of ANTERION and the reference device
Repeatability and Reproducibility 4 | 1 day
  Reproducibility and repeatability of Anterior Segment Angles parameter [°] of ANTERION and the reference device
Repeatability and Reproducibility 5 | 1 day
  Reproducibility and repeatability of TISA parameters [mm2] of ANTERION and the reference device
Repeatability and Reproducibility 6 | 1 day
  Reproducibility and repeatability of AOD parameters [µm] of ANTERION and the reference device
Agreement 1 | 1 day
  Agreement of Spur to Spur distance parameter [mm] between the ANTERION and the reference device
Agreement 2 | 1 day
  Agreement of Angle to Angle distance parameter [mm] between the ANTERION and the reference device
Agreement 3 | 1 day
  Agreement of Lens Vault parameter [µm] between the ANTERION and the reference device
Agreement 4 | 1 day
  Agreement of Anterior Segment Angles parameter [°] between the ANTERION and the reference device
Agreement 5 | 1 day
  Agreement of TISA parameters [mm2] between the ANTERION and the reference device
Agreement 6 | 1 day
  Agreement of AOD parameters [µm] between the ANTERION and the reference device

SECONDARY OUTCOMES:
Adverse Events Rate | 1 day
  Adverse events found during the clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Dul, Principal Investigator — State University of New York College of Optometry
Locations (1):
- State University of New York College of Optometry, New York, New York, United States